CLINICAL TRIAL: NCT03804190
Title: Work-Related Musculoskeletal Disorders Among Egyptian Otorhinolarngologist
Brief Title: Work-Related Musculoskeletal Disorders Among Otorhinolarngologists
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, HAhmed, assistant professor, Cairo University
Other Study IDs: NO:P.T.REC/012/002090
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-12

CONDITIONS: Work-Related Musculoskeletal Disorders Among EGYPTIAN Otorhinolarngologists

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1-5years experience: 1-5years of experience working as otorhinolaryngologist
  Interventions: Other: questionaire
- 5-10 years experience: 5-10years of experience working as otorhinolaryngologist
  Interventions: Other: questionaire
- 10-15years experince: 10-15years of experience working as otorhinolaryngologist
  Interventions: Other: questionaire
- 15_20years experience: 15-20years of experience working as otorhinolaryngologist
  Interventions: Other: questionaire

INTERVENTIONS:
Other: questionaire — dutch musculoskeletal questionaire

SUMMARY:
Work-Related Musculoskeletal Disorders Among Otorhinolarngologists

DETAILED DESCRIPTION:
Musculoskeletal disorders(MSD) are one of the most common causes of occupational injuries and disability in industrialized nations and developing countries .with substantial financial consequences due to workers' compensation and medical expenses Otolaryngology (pronounced oh/toe/lair/in/goll/oh/jee) is the oldest medical specialty in the United States. Otolaryngologists are physicians trained in the medical and surgical management and treatment of patients with diseases and disorders of the ear, nose, throat (ENT), and related structures of the head and neck. They are commonly referred to as ENT physicians.

MSD were identified as a significant issue for the profession and Research has recognized that MSD in Otolaryngology contribute considerably to sick leave, reduced productivity and leaving the profession Because there are few studies available about MSD among Egyptian otolaryngologists So, the purpose of this study is to investigate musculoskeletal disorders among Egyptian otorhinlaryngologist and the relationship between the risk factors and the development of musculoskeletal disorders among Egyptian otolaryngologists

ELIGIBILITY:
Inclusion Criteria:

- otorhinolaryngologist in cairo university hospitals ,cairo teaching hospitasl will participate in the study.

1. General and specialized otolaryngologists will be included in the study.
2. Both genders will be included in the study.
3. 1-20 years of experience.

Exclusion Criteria:

* Otorhinologist will be excluded if :

  1. they had musculoskeletal abnormalities due to other causes not work related (i.e. congenital,traumatic,neurological).
  2. They had any systemic diseases such as uncontrolled diabetes, which may influence the musculoskeletal system
  3. Otolaryngologists with previous operation involving locomotors system.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: otorhinolaryngologist in cairo university hospitals ,cairo teaching hospitasl will participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
prevelance of work related musculoskeletal disorders among otorhinolaryngologist and work related musculoskeletal disorders among otorhinolaryngologist | one year
  work related musculoskeletal disorders among otorhinolaryngologist

CONTACTS AND LOCATIONS:
Overall Officials: daoo ibrahim, assistant professor, Study Director — Cairo University; hamada ahmed, lecterur, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided